CLINICAL TRIAL: NCT03926117
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate Reduction in Inflammation in Patients With Advanced Chronic Renal Disease Utilizing Antibody Mediated IL-6 Inhibition
Brief Title: Trial to Evaluate Reduction in Inflammation in Patients With Advanced Chronic Renal Disease Utilizing Antibody Mediated IL-6 Inhibition
Acronym: RESCUE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN6018-4779
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases; Inflammation
Keywords: IL-6; CRP; Chronic Kidney Disease; Cardiovascular Disease; Inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Inflammation; Cardiovascular Diseases | interventions — ziltivekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Biological: Ziltivekimab
- Ziltivekimab 7.5 mg (Experimental)
  Interventions: Biological: Ziltivekimab
- Ziltivekimab 15 mg (Experimental)
  Interventions: Biological: Ziltivekimab
- Ziltivekimab 30 mg (Experimental)
  Interventions: Biological: Ziltivekimab

INTERVENTIONS:
Biological: Ziltivekimab — human IgG1k anti-human IL-6 monoclonal antibody
  Other Names: COR-001

SUMMARY:
Patients with chronic kidney disease, who have evidence of systemic inflammation with increased cardiovascular risk, will be enrolled into this trial. The purpose of this trial is to determine a dose to select for a potential cardiovascular outcome trial with Ziltivekimab. Doses to be tested will be 7.5 mg, 15 mg and 30 mg subcutaneous monthly compared to placebo for six months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Stage 3-5 CKD
* hs-CRP > 2.0 mg/L
* Comply with contraception

Exclusion Criteria:

* Low neutrophil count
* Low platelet count
* Spot urine protein to creatinine ration > 4000 mg/g
* ALT/AST >2.5x ULN
* TSAT < 10%
* Positive TB test
* Evidence of HIV, hepatitis B
* Blind or illiterate
* Expected to require blood transfusion
* Thromboembolic event within 12-weeks
* Evidence of active infection
* Peptic ulcer disease, diverticulitis, inflammatory bowel disease
* Uncontrolled hypertension
* Planned coronary revascularization
* Major cardiac surgery, CHF
* Active malignancy, bone marrow or organ transplant
* Allergy to study drug
* Treatment with investigational drug, treatment with HIF stabilizer or ESA
* Use of immunosuppressive drugs, systemic antibiotics
* Breastfeeding, any other significant medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (49):
- United States (49):
  - Central Alabama Research, Birmingham, Alabama
  - Aventiv Research, Mesa, Arizona
  - Arizona Kidney Disease and Hypertension Center, Phoenix, Arizona
  - Elite Clinical Studies, Phoenix, Arizona
  - North America Research Institute, Lynwood, California
  - North America Research Institute, Riverside, California
  - Apex Research of Riverside, Riverside, California
  - North America Research Institute, San Dimas, California
  - Western Nephrology and Metabolic Bone Disease, PC, Arvada, Colorado
  - AMPM Research Clinic, Miami, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - Florida Premier Research Institue, LLC, Winter Park, Florida
  - Southeastern Clinical Research Institute, LLC, Augusta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Investigator Research by Design, LLC, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Clinical Trials of America, LLC - West Monroe, Monroe, Louisiana
  - Capital Nephrology, Greenbelt, Maryland
  - Onyx Clinical Research, Caro, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - St. Clair Nephrology Research, Roseville, Michigan
  - Nephrology Research of Michigan, Saint Clair Shores, Michigan
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Julia and Israel Waldbaum Dialysis Center, Great Neck, New York
  - Northport VAMC, Northport, New York
  - DaVita Clinical Research, The Bronx, New York
  - Mountain Kidney and Hypertension Associates, Asheville, North Carolina
  - Metrolina Nephrology Associates, PA, Charlotte, North Carolina
  - Metrolina Nephrology Associates, Charlotte, North Carolina
  - Southeastern Nephrology - Whiteville, Whiteville, North Carolina
  - Southeastern Nephrology Associates - Wilmington, Wilmington, North Carolina
  - Summit Research Group, LLC, Stow, Ohio
  - Northeast Clinical Research Center, Allentown, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Piedmont Research Partners, LLC, Fort Mill, South Carolina
  - Mountain View CLinical Research - Greer, Greer, South Carolina
  - Knoxville Kidney Center, PLLC, Knoxville, Tennessee
  - Nephrology Associates, PC, Nashville, Tennessee
  - Renal Disease Research Institute, Dallas, Texas
  - Vilo Research Group, Inc, Houston, Texas
  - Biopharma Informatick Inc. Research Center, Houston, Texas
  - Juno Research, LLC - Northwest, Houston, Texas
  - North Hills Medical Research, Inc, North Richland Hills, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - San Antonio Kidney Disease Center Physicians Group, PLLC, San Antonio, Texas
  - University of Vermont, Burlington, Vermont
  - Southside Urology and Nephrology, Danville, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Clinical Investigation Specialist, Inc, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Kreiner FF, Kraaijenhof JM, von Herrath M, Hovingh GKK, von Scholten BJ. Interleukin 6 in diabetes, chronic kidney disease, and cardiovascular disease: mechanisms and therapeutic perspectives. Expert Rev Clin Immunol. 2022 Apr;18(4):377-389. doi: 10.1080/1744666X.2022.2045952. Epub 2022 Mar 1. PMID 35212585
- [Derived] Aherrahrou R, Reinberger T, Hashmi S, Erdmann J. GWAS breakthroughs: mapping the journey from one locus to 393 significant coronary artery disease associations. Cardiovasc Res. 2024 Nov 5;120(13):1508-1530. doi: 10.1093/cvr/cvae161. PMID 39073758
- [Derived] Pergola PE, Davidson M, Jensen C, Mohseni Zonoozi AA, Raj DS, Andreas Schytz P, Tuttle KR, Perkovic V. Effect of Ziltivekimab on Determinants of Hemoglobin in Patients with CKD Stage 3-5: An Analysis of a Randomized Trial (RESCUE). J Am Soc Nephrol. 2024 Jan 1;35(1):74-84. doi: 10.1681/ASN.0000000000000245. Epub 2023 Dec 13. PMID 38088558
- [Derived] Ridker PM, Devalaraja M, Baeres FMM, Engelmann MDM, Hovingh GK, Ivkovic M, Lo L, Kling D, Pergola P, Raj D, Libby P, Davidson M; RESCUE Investigators. IL-6 inhibition with ziltivekimab in patients at high atherosclerotic risk (RESCUE): a double-blind, randomised, placebo-controlled, phase 2 trial. Lancet. 2021 May 29;397(10289):2060-2069. doi: 10.1016/S0140-6736(21)00520-1. Epub 2021 May 17. PMID 34015342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 52 clinical sites in the United States.
Pre-assignment Details: Participants were randomized 1:1:1:1 to one of three Ziltivekimab dose levels (7.5 milligram (mg), 15 mg, or 30 mg) or matching placebo.
Groups:
- Placebo: Participants received subcutaneous (SC) injection of placebo matched to Ziltivekimab once in every 28 days at weeks 1, 5, 9, 13, 17 and 21. Participants were followed up for safety from week 25 through week 32.
- Ziltivekimab 7.5 mg: Participants received SC injection of 7.5 mg Ziltivekimab once in every 28 days at weeks 1, 5, 9, 13, 17 and 21. Participants were followed up for safety from week 25 through week 32.
- Ziltivekimab 15 mg: Participants received SC injection of 15 mg Ziltivekimab once in every 28 days at weeks 1, 5, 9, 13, 17 and 21. Participants were followed up for safety from week 25 through week 32.
- Ziltivekimab 30 mg: Participants received SC injection of 30 mg Ziltivekimab once in every 28 days at weeks 1, 5, 9, 13, 17 and 21. Participants were followed up for safety from week 25 through week 32.
Period: Overall Study
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Started | 66 | 66 | 66 | 66
Intent-to-treat Analysis Population | 66 | 66 | 66 | 66
Safety Analysis Population | 65 | 65 | 66 | 65
Treated | 65 | 65 | 66 | 65
Completed | 60 | 57 | 60 | 59
Not Completed | 6 | 9 | 6 | 7
Not completed — Unclassified | 1 | 4 | 1 | 4
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0
Not completed — Adverse Event | 1 | 2 | 3 | 1
Not completed — Randomized but not treated | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg | Total
Number analyzed (Participants) | 66 | 66 | 66 | 66 | 264
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (10.81) | 67.2 (10.67) | 65.9 (9.42) | 67.1 (10.55) | 66.4 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 36 | 32 | 129
  Male | 37 | 34 | 30 | 34 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 12 | 15 | 19 | 71
  Not Hispanic or Latino | 41 | 54 | 51 | 46 | 192
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 50 | 48 | 49 | 52 | 199
  Race: Black or African American | 16 | 18 | 12 | 14 | 60
  Race: Asian | 0 | 0 | 3 | 0 | 3
  Race: Native Hawaiian or other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Race: Other | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in High-sensitivity C-reactive Protein (Hs-CRP) Levels
Description: Percent change from baseline in hs-CRP levels at week 13 are presented.
Time Frame: Baseline (average of the hs-CRP value prior to randomization and day 1), week 13
Population: ITT analysis population included all randomized participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 57 | 58 | 61 | 57
Percent change | -4.49 [-35.54 to 46.27] | -76.57 [-86.89 to -57.14] | -88.12 [-92.11 to -78.95] | -91.64 [-95.19 to -86.15]
Statistical Analysis 1: Comparison: Placebo vs Ziltivekimab 7.5 mg; Percent change from baseline is analyzed using nonparametric Hodges-Lehmann estimator. The nonparametric analysis accounts for covariates baseline hemoglobin (greater than or equal to (>=) 11 or less than (<) 11 grams per deciliter (g/dL)) and chronic kidney disease stage (3, 4 or 5) by aligning responses within each stratum defined by the covariates prior to analysis; Test type: Superiority; p < 0.0001, Hodges-Lehmann method; Median Difference (Final Values) = -66.20, 95% CI 2-sided [-86.15 to -49.12]
Statistical Analysis 2: Comparison: Placebo vs Ziltivekimab 15 mg; Percent change from baseline is analyzed using nonparametric Hodges-Lehmann estimator. The nonparametric analysis accounts for covariates baseline hemoglobin (>= 11 or < 11 g/dL) and chronic kidney disease stage (3, 4 or 5) by aligning responses within each stratum defined by the covariates prior to analysis; Test type: Superiority; p < 0.0001, Hodges-Lehmann method; Median Difference (Final Values) = -77.71, 95% CI 2-sided [-94.98 to -62.97]
Statistical Analysis 3: Comparison: Placebo vs Ziltivekimab 30 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Hodges-Lehmann method; Median Difference (Final Values) = -87.76, 95% CI 2-sided [-101.00 to -70.54]

2. Secondary Outcome: Percent Change From Baseline in Serum Amyloid A (SAA)
Description: Percent change from baseline in SAA at week 13 are presented.
Time Frame: Baseline (average of the values at week -1 and day 1), week 13
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 57 | 58 | 60 | 56
Percent change | 1.82 [-18.42 to 50.98] | -40.24 [-61.54 to -12.38] | -49.80 [-63.90 to -31.54] | -42.45 [-68.91 to -13.48]

3. Secondary Outcome: Percent Change From Baseline in Fibrinogen
Description: Percent change from baseline in fibrinogen at week 13 are presented.
Time Frame: Baseline (day 1), week 13
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 55 | 55 | 60 | 54
Percent change | -1.62 [-12.90 to 13.35] | -25.20 [-33.27 to -7.93] | -24.69 [-36.25 to -16.48] | -37.17 [-44.94 to -28.57]

4. Secondary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious AEs (TESAEs), Severe Hematologic AEs, Severe Non-hematologic AEs, and AEs Leading to Drug Discontinuation
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. TEAEs are defined as AEs that initiated or worsened on or after the date of first dose of study drug up to the end of safety-follow-up. A SAE was defined as any untoward medical occurrence that at any dose results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization results in persistent or significant disability/incapacity, or may have caused a congenital anomaly/birth defect, or requires intervention to prevent permanent impairment or damage. TEAEs that met any of these criteria were considered severe hematologic AEs: grade 3 neutropenia, grade 3 anemia, grade 3 leukopenia, grade 3 lymphopenia, grade 3 eosinophilia, and grade 3 thrombocytopenia.
Time Frame: From week 0 to week 32
Population: The safety analysis population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 65 | 65 | 66 | 65
Percentage of participants
  TEAEs | 69.2 | 66.2 | 66.7 | 72.3
  TESAEs | 15.4 | 20.0 | 13.6 | 12.3
  Severe hematologic AEs | 1.5 | 0.0 | 1.5 | 0.0
  Severe non-hematologic AEs | 10.8 | 18.5 | 9.1 | 12.3
  AEs leading to study drug discontinuation | 4.6 | 6.2 | 7.6 | 4.6

5. Secondary Outcome: Percentage of Participants With Thrombolysis in Myocardial Infarction (TIMI) Major Bleeding Events
Description: Bleeding events were classified using the TIMI bleeding classification as follows: 1) major: intracranial hemorrhage or a >=5 g/dL decrease in the hemoglobin concentration or a >=15 percent (%) absolute decrease in the hematocrit; 2) minor: (a) observed blood loss: >=3 g/dL decrease in the hemoglobin concentration or >=10% decrease in the hematocrit. (b) no observed blood loss: >=4 g/dL decrease in the hemoglobin concentration or >=12% decrease in the hematocrit; 3) minimal: any clinically overt sign of hemorrhage (including imaging) that was associated with a < 3 g/dL decrease in the hemoglobin concentration or <9% decrease in the hematocrit.
Time Frame: From week 0 to week 32
Population: The safety analysis population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 65 | 65 | 66 | 65
Percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

6. Secondary Outcome: Percentage of Participants With Any Treatment-emergent Adverse Events of Special Interest (AESI)
Description: An AE was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. AESI included serious infections, malignancies, anaphylaxis occurring at any time, even if considered unrelated to the study drug, gastrointestinal perforations, hypersensitivity reaction during investigational product (IP) administration, neutrophils per cubic millimeter (500/mm^3) (severe) or neutrophils <1000/mm^3 (severe) with evidence of concurrent infection, severe injection-related reactions, thrombocytopenia (platelet count <50,000/mm^3 (severe)) or platelet count <75,000/mm^3 (moderate) with evidence of concurrent TIMI major bleeding.
Time Frame: From week 0 to week 32
Population: The safety analysis population included all randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 65 | 65 | 66 | 65
Percentage of participants
  Serious infection | 4.6 | 10.8 | 4.5 | 3.1
  Malignancy | 1.5 | 0.0 | 1.5 | 1.5
  Anaphylaxis | 0.0 | 0.0 | 0.0 | 0.0
  Gastrointestinal perforations | 0.0 | 0.0 | 0.0 | 0.0
  Hypersensitivity reaction during IP administration | 0.0 | 0.0 | 0.0 | 0.0
  Neutropenia, severe | 0.0 | 0.0 | 0.0 | 0.0
  Neutropenia, severe with evidence of concurrent infection | 0.0 | 0.0 | 0.0 | 0.0
  Severe injection-related reaction | 0.0 | 0.0 | 0.0 | 0.0
  Thrombocytopenia, moderate with evidence of concurrent TIMI major bleeding | 0.0 | 0.0 | 0.0 | 0.0
  Thrombocytopenia, severe | 0.0 | 0.0 | 0.0 | 0.0

7. Secondary Outcome: Change in Systolic Blood Pressure (SBP)
Description: Change from baseline in systolic blood pressure at week 32 are presented.
Time Frame: Baseline (week 1), week 32
Population: The safety analysis population included all randomized participants who received at least 1 dose of study drug. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 52 | 52 | 55 | 53
Millimeters of mercury (mmHg) | 4.8 (15.94) | 4.9 (16.31) | 0.6 (18.89) | 1.2 (14.71)

8. Secondary Outcome: Change in Diastolic Blood Pressure (DBP)
Description: Change from baseline in diastolic blood pressure at week 32 are presented.
Time Frame: Baseline (week 1), week 32
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 52 | 52 | 55 | 53
mmHg | 0.7 (10.33) | 2.9 (10.97) | 1.1 (11.17) | 3.1 (10.35)

9. Secondary Outcome: Change in Respiratory Rate
Description: Change from baseline in respiratory rate at week 32 are presented.
Time Frame: Baseline (week 1), week 32
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Breaths per minute (breaths/min)
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 52 | 52 | 55 | 53
Breaths per minute (breaths/min) | 0.4 (2.24) | 0.2 (2.18) | -0.7 (2.36) | -0.5 (1.62)

10. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change from baseline in BMI at week 24 are presented.
Time Frame: Baseline (week 1), week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Kilograms per square meter (kg/m^2)
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 32 | 31 | 34 | 30
Kilograms per square meter (kg/m^2) | 0.13 (1.102) | 0.51 (1.904) | 0.58 (1.664) | 0.40 (0.879)

11. Secondary Outcome: Change in Heart Rate
Description: Change from baseline in heart rate at Week 32 are presented.
Time Frame: Baseline (week 1), week 32
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 52 | 52 | 55 | 53
Beats per minute (beats/min) | 2.8 (9.70) | 1.5 (10.18) | -0.6 (8.93) | 1.2 (11.56)

12. Secondary Outcome: Change in Temperature
Description: Change from baseline in temperature at week 32 are presented.
Time Frame: Baseline (week 1), week 32
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Degree Celsius (°C)
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 52 | 52 | 55 | 53
Degree Celsius (°C) | 0.03 (0.456) | -0.01 (0.430) | -1.13 (8.366) | -0.02 (0.615)

13. Secondary Outcome: Change in Electrocardiogram (ECG)
Description: The ECG was assessed by the investigator at baseline (week -1) and week 24 and categorised as abnormal clinically significant, abnormal not clinically significant, indeterminate, normal, not evaluable and unknown. Number of participants in each ECG category at baseline and week 24 are presented.
Time Frame: Baseline (week -1), Week 24
Population: The safety analysis population included all randomized participants who received at least 1 dose of study drug. 'Overall Number of Participants Analyzed' = participants with available data and 'Number Analyzed' = number of participants with available data for each category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 65 | 65 | 65 | 64
Participants
  Baseline (week-1): Abnormal, clinically significant | 0 | 0 | 0 | 0
  Baseline (week-1): Abnormal, not clinically significant | 44 | 38 | 40 | 46
  Baseline (week-1): Indeterminate | 0 | 0 | 0 | 0
  Baseline (week-1): Normal | 21 | 27 | 25 | 18
  Baseline (week-1): Not evaluable | 0 | 0 | 0 | 0
  Baseline (week-1): Unknown | 0 | 0 | 0 | 0
  Week 24: number analyzed (Participants) | 50 | 54 | 53 | 52
  Week 24: Abnormal, clinically significant | 0 | 0 | 0 | 0
  Week 24: Abnormal, not clinically significant | 36 | 32 | 35 | 34
  Week 24: Indeterminate | 0 | 0 | 0 | 0
  Week 24: Normal | 14 | 22 | 18 | 18
  Week 24: Not evaluable | 0 | 0 | 0 | 0
  Week 24: Unknown | 0 | 0 | 0 | 0

14. Secondary Outcome: Change in Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AAT) Levels
Description: Change from baseline in ALP, ALT and AAT levels at week 32 are presented.
Time Frame: Baseline (week 1), week 32
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 52 | 53 | 55 | 53
Units per liter (U/L)
  ALP: Change from baseline to Week 32 | -1.9 (14.75) | -6.3 (18.28) | -9.6 (18.56) | -15.7 (13.94)
  ALT: Change from baseline to Week 32 | 1.3 (5.53) | 2.6 (6.56) | 5.3 (11.76) | 7.2 (13.73)
  AAT: Change from baseline to Week 32 | 0.6 (6.05) | 2.3 (4.65) | 3.3 (8.28) | 4.8 (9.15)

15. Secondary Outcome: Change in Bicarbonate, Chloride, Potassium, Sodium
Description: Change from baseline in bicarbonate, chloride, potassium, sodium at week 32 are presented.
Time Frame: Baseline (week 1), week 32
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 52 | 53 | 55 | 53
millimoles per liter (mmol/L)
  Bicarbonate: Change from baseline to Week 32 | -0.9 (2.60) | -0.3 (2.66) | -0.7 (2.96) | -1.2 (2.72)
  Chloride: Change from baseline to Week 32 | 1.7 (3.86) | 0.0 (3.27) | 0.7 (2.95) | 0.9 (3.39)
  Potassium: Change from baseline to Week 32 | 0.00 (0.445) | -0.28 (0.739) | -0.29 (0.570) | -0.16 (0.567)
  Sodium: Change from baseline to Week 32 | 1.0 (2.92) | 0.0 (2.70) | 0.3 (2.44) | -0.1 (2.20)

16. Secondary Outcome: Change in Direct Bilirubin, Bilirubin, Calcium, Creatinine, Glucose, Phosphate and Urea Nitrogen
Description: Change from baseline in direct bilirubin, bilirubin, calcium, creatinine, glucose, phosphate and urea nitrogen at week 32 are presented.
Time Frame: Baseline (week 1), week 32
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 52 | 53 | 55 | 53
milligrams per deciliter (mg/dL)
  Direct Bilirubin: Change from baseline to Week 32 | -0.007 (0.0297) | 0.008 (0.0263) | 0.018 (0.0300) | 0.009 (0.0367)
  Bilirubin: Change from baseline to Week 32 | -0.028 (0.1284) | 0.060 (0.1013) | 0.105 (0.1576) | 0.065 (0.1812)
  Calcium: Change from baseline to Week 32 | -0.04 (0.494) | 0.09 (0.407) | 0.16 (0.524) | 0.11 (0.405)
  Creatinine: Change from baseline to Week 32 | -0.041 (0.6114) | 0.216 (0.5291) | 0.054 (0.3404) | 0.141 (0.4618)
  Glucose: Change from baseline to Week 32 | -15.1 (83.48) | 8.9 (80.50) | 9.2 (64.86) | 1.7 (48.43)
  Phosphate: Change from baseline to Week 32 | -0.04 (0.778) | 0.04 (0.766) | 0.02 (0.620) | 0.21 (0.641)
  Urea Nitrogen: Change from baseline to Week 32 | 0.4 (11.76) | 4.7 (12.15) | 1.6 (7.97) | 5.6 (13.89)

17. Secondary Outcome: Follicle Stimulating Hormone (FSH) Levels
Description: FSH levels at baseline (week -1) are presented.
Time Frame: Baseline (week -1)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 8 | 15 | 16 | 13
International units per liter (IU/L) | 57.45 (20.496) | 72.70 (36.519) | 77.49 (33.827) | 58.79 (48.167)

18. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADAs)
Description: Participants who had at least 1 positive sample (treatment-boosted or treatment-induced) at any time after their first Ziltivekimab administration were classified as positive for ADAs. In the instance that a participant had a positive sample at the baseline visit, the participant was considered positive only if the peak titer of the post-treatment sample was at least 2-fold higher (i.e., >=2-fold) than the titer of the baseline sample. Number of participants positive for antibodies to Ziltivekimab are presented.
Time Frame: From week 0 to week 32
Population: Analysis population included all randomized participants. 'Overall Number of Participants Analyzed' = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
Number analyzed (Participants) | 65 | 65 | 66 | 64
Participants | 0 | 4 | 5 | 7

ADVERSE EVENTS:
Time Frame: From week 0 to week 32
Description: All presented AEs are treatment-emergent adverse events (TEAEs). A TEAE was defined as an AE that initiated or worsened on or after the date of first dose of study drug up to the end of the safety follow-up (week 32). The results are based on the safety analysis set which included all randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | Ziltivekimab 7.5 mg | Ziltivekimab 15 mg | Ziltivekimab 30 mg
All-Cause Mortality (participants affected / at risk) | 1/65 | 0/65 | 0/66 | 0/65
Serious Adverse Events (participants affected / at risk) | 10/65 | 13/65 | 9/66 | 8/65
Other Adverse Events (participants affected / at risk) | 19/65 | 22/65 | 18/66 | 17/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | Ziltivekimab 7.5 mg (N=65) | Ziltivekimab 15 mg (N=66) | Ziltivekimab 30 mg (N=65)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous graft site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | Ziltivekimab 7.5 mg (N=65) | Ziltivekimab 15 mg (N=66) | Ziltivekimab 30 mg (N=65)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 2 (2) | 1 (1) | 3 (3)
Dizziness (Nervous system disorders) | 1 (2) | 3 (3) | 4 (4) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 5 (6) | 6 (6) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (3) | 4 (5) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 3 (3) | 3 (3)
Oedema peripheral (General disorders) | 2 (3) | 4 (4) | 1 (1) | 4 (5)
Urinary tract infection (Infections and infestations) | 4 (5) | 4 (4) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT03926117/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03926117/SAP_001.pdf